CLINICAL TRIAL: NCT03272139
Title: Interscalene Block Versus Superior Trunk Block: A Randomized Controlled Clinical Trial
Brief Title: Interscalene Block Versus Superior Trunk Block
Acronym: STB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-0979
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Joint Disease; Pain; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Joint Diseases; Pain; Acute Pain; Chronic Pain | interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- interscalene block (ISB) (Experimental): The interscalene block will be done using an ultrasound-guided, in-plane approach. The anesthesiologists will target below the C5 nerve root. A 22 gauge 1.5-2 inch needle is advanced in-plane from lateral to medial through the middle scalene muscle until the needle tip is positioned in the interscalene groove between the C5 and C6 nerve roots. 15 20 ml of 0.5% bupivacaine will be injected.
  Interventions: Drug: Bupivacaine; Device: Ultrasound
- superior trunk block (STB) (Experimental): The superior trunk block will be performed at the point immediately distal to the roots when the c5-c6 form the superior trunk and lies anterior to the middle scalene muscle and below the deep cervical fascia, before the suprascapular nerve arises and goes into the omohyoid. A 22g 1.5-2inch needle will be advanced in-plane from lateral to medial. The needle tip will be placed lateral to the superior trunk and 15 20 ml of 0.5% bupivacaine will be injected just inferior to the deep cervical fasica. Local circumferential spread will be achieved both anterior and posterior to the superior trunk.
  Interventions: Drug: Bupivacaine; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacaine — Anesthetic that will help treat pain and sensation after shoulder arthroscopy
Device: Ultrasound — Ultrasound will help guide the anesthesiologist in performing the different nerve blocks

SUMMARY:
Sparing the phrenic nerve by administering ultrasound-guided low volume superior trunk block (STB) and interscalene block (ISB) for arthroscopic shoulder surgery (labral repair, stabilization, rotator cuff repair).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be undergoing primary unilateral labral repair/stabilization of the shoulder
* Age 18 to 80 years
* Planned use of general anesthesia with LMA and interscalene or superior trunk block
* Ability to follow study protocol
* English speaking
* ASA I - III

Exclusion Criteria:

Pre-existing neuropathy of the operative limb

* Younger than 18 years old and older than 80
* Patients with pulmonary severe respiratory disease
* Allergy to one of the study medications
* Chronic gabapentin/pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Contraindication to general anesthesia, interscalene or superior trunk block
* Herniated Cervical Disk, Cervical Myelopathy
* BMI >35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interscalene Block (ISB) | Superior Trunk Block (STB)
Started | 63 | 63
Completed | 63 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interscalene Block (ISB) | Superior Trunk Block (STB) | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.0 [38.0 to 59.0] | 51.5 [37.0 to 60.0] | 51 [37 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 44 | 49 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 4 | 8
  White | 52 | 54 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.8 [24.4 to 29.6] | 27.2 [24.8 to 29.8] | 26.8 [24.8 to 29.8]
Length of Surgery [Median (Inter-Quartile Range); unit: minutes] | 46.0 [35.0 to 66.0] | 49.0 [32.0 to 62.0] | 48 [33 to 63]
ASA Class [Number; unit: participants] — ASA Classification System is to assess and communicate a patient's pre-anesthesia medical co-morbidities. ASA1 is a normal healthy patient. ASA2 is a patient with mild systemic disease and ASA3 is a patient with severe systemic disease.
  participants
    ASA 1 | 18 | 10 | 28
    ASA 2 | 44 | 52 | 96
    ASA 3 | 1 | 1 | 2
Laterality [Number; unit: participants]
  LEFT Shoulder Arthroscopy | 28 | 23 | 51
  Right Shoulder Arthroscopy | 35 | 40 | 75
Baseline NRS [Median (Inter-Quartile Range); unit: units on a scale] — Numerical Rating Scale 0-10; with 0 being no pain and 10 pain as bad as you can imagine.
  units on a scale | 2.0 [0 to 3.0] | 2.0 [0 to 3.0] | 2.0 [0 to 3.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Hemidiaphragmatic Paralysis (HDP)
Description: Our primary outcome will be the incidence of hemidiaphragmatic paralysis (HDP) with superior trunk block and interscalene blocks as measured by ultrasound before and after the surgery.
Time Frame: Day of Surgery, diagnosis confirmed from trained anesthesiologist ultrasound readers
Measure: Number; unit: participants
Arm/Group | Interscalene Block (ISB) | Superior Trunk Block (STB)
Number analyzed (Participants) | 63 | 62
participants
  HDP | 45 | 3
  No HDP | 18 | 59

2. Primary Outcome: Numerical Pain Rating System (NRS) Pain Scores
Description: Numerical Pain Rating System Pain scores after the superior trunk block and interscalene block at rest measured after the surgery every 30 minute until discharge according to the Post Anaesthetic Discharge Scoring System.
  Numerical Rating Scale 0-10; with 0 being no pain and 10 pain as bad as you can imagine.
Time Frame: Average pain scores at rest recorded Day of Surgery every 30 minutes until discharge according to Post Anaesthetic Discharge Scoring System
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Interscalene Block (ISB) | Superior Trunk Block (STB)
Number analyzed (Participants) | 63 | 62
units on a scale | 0 [0 to 2] | 0 [0 to 3]

3. Secondary Outcome: Block Duration
Description: Length of nerve block reported by Phone call on POD 1 and POD 2 by patient phone call
Time Frame: Time of block wearing off recorded on Post Operative Day 1 and Post Operative Day 2 as reported via patient phone call.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Interscalene Block (ISB) | Superior Trunk Block (STB)
Number analyzed (Participants) | 57 | 61
Hours | 23.18 [19.95 to 25.53] | 23.15 [19.12 to 30.07]

ADVERSE EVENTS:
Time Frame: From Post Op Day 1 to Post Op Day 7
Description: Incidence of paresthesia / neuropraxia ( POD1, POD ): persistent tingling, numbness in POD1, if patient reports persistent neuropraxia after POD2, will follow up on POD7. If persists, will notify attending anesthesiologist and continue to follow until postoperative neurologic symptoms (PONS) resolves.
Arm/Group | Interscalene Block (ISB) | Superior Trunk Block (STB)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT03272139/Prot_SAP_000.pdf